CLINICAL TRIAL: NCT01111370
Title: Effectiveness and Safety Study of the DexCom™ G4 Continuous Glucose Monitoring System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PTL900360
Record Dates: First submitted 2010-04-22; First posted 2010-04-27 (Estimated); Results first posted 2017-03-27 (Actual); Last update posted 2017-03-27 (Actual); Status verified 2015-08

CONDITIONS: Diabetes Mellitus
Keywords: diabetes mellitus requiring insulin
MeSH Terms: conditions — Diabetes Mellitus | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CGM (Experimental): continuous glucose monitoring system
  Interventions: Device: DexCom™ G4 Continuous Glucose Monitoring System

INTERVENTIONS:
Device: DexCom™ G4 Continuous Glucose Monitoring System — Continuous Glucose Monitoring System
  Other Names: Continuous Glucose Monitoring System

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the G4 System when worn for up to 7-days by subjects >18 years-old with diabetes mellitus requiring insulin.

Device performance will be primarily evaluated in terms of the proportion of G4 System values that are within ±20% of YSI reference value for glucose levels >80 mg/dL and ±20 mg/dL at meter glucose levels <80 mg/dL. These G4-YSI matched pairs will be collected during in-clinic sessions on Days 1, 4, and 7 of Sensor wear. The proportion of matched pairs from this study (PTL-900360) meeting the above criteria will be compared to the proportion of such points observed in the DexCom clinical study that supported approval of the SEVEN PLUS System (PTL 300012).

Safety data of the G4 System will also be collected and safety will be characterized by the incidence of Adverse Device Effects, Serious Adverse Device Events, and Unanticipated Adverse Device Effects experienced by study participants.

DETAILED DESCRIPTION:
This will be a non-randomized, single-armed study conducted in the United States. Following screening, a minimum of 60 to a maximum of 80 subjects at up to 4 clinical sites will be enrolled. All participants will wear the G4 Sensor for one 7-day wear period (~168 hours). A subset of 20-30 subjects will wear two G4 Systems (one of which will be blinded) during the 7-day wear period for the purposes of assessing precision. During home use, subjects will be asked to use the meter provided to them to take fingersticks for calibration and diabetes management. Subjects will also be asked to confirm high and low G4 System glucose alerts/alarms by taking a comparative fingerstick immediately after receiving an alert/alarm.

All subjects will participate in one, 8-hour in-clinic session on Day 1, 4, or 7 of the study to collect accuracy information against a laboratory standard (YSI) and against SMBG. During the in-clinic session, subjects will have venous blood draws for evaluation of the YSI blood glucose measurements. Carbohydrate consumption and insulin dosing may be manipulated during the in-clinic session to ensure a wide range of glucose values. For the duration of this study, subjects will be instructed to use G4 System information as an adjunct to (and not as a replacement for) standard SMBG guidance of diabetes self-management.

Subjects will perform G4 Sensor insertions at the clinic under supervision of study staff. Sensor insertion sites will be examined after removal of the Sensor(s). Study staff will document any irritation and/or Adverse Device Effects.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older;
2. Have been diagnosed with insulin-requiring diabetes and are on multiple daily injections (MDI) or Continuous Subcutaneous Insulin Infusion (CSII) insulin therapy;
3. Willing not to inject insulin or wear an insulin pump insertion set within 3 inches from the Sensor site during Sensor wear;
4. Willing to use only the blood glucose meter provided to them for self-monitoring of blood glucose (SMBG) during Sensor wear;
5. Willing to participate in one, 8-hour in-clinic session and be willing to take 4 fingersticks per hour and have 4 blood draws per hour for the entire 8-hour duration;
6. Willing to take a minimum of 6 fingersticks per day during home use (2 for calibration purposes, 4 for comparative purposes);
7. Willing to refrain from the use of acetaminophen during the Sensor insertion period and for at least 24-hours prior to Sensor insertion;
8. Willing not to schedule a magnetic resonance (MRI) scan, computed tomography (CT) scan, or x-ray, for the duration of the study;
9. Able to speak, read, and write English.

Exclusion Criteria:

1. Have extensive skin changes/diseases that preclude wearing the Sensor on normal skin (e.g. extensive psoriasis, recent burns or severe sunburn, extensive eczema, extensive scarring, extensive tattoos, dermatitis herpetiformis) at the proposed wear sites;
2. Subjects who have a known allergy to medical-grade adhesives;
3. Are pregnant as demonstrated by a positive pregnancy test within 72 hours of insertion;
4. Have a hematocrit that is less than 30%, or greater than 55%;
5. Current participation in another investigational study protocol (if a subject has recently completed participation in another drug study, the subject must have completed that study at least 30 days prior to being enrolled in this study);
6. Have any condition that, in the opinion of the Investigator, would interfere with their participation in the trial or pose an excessive risk to study staff handling venous blood samples (e.g., known history of hepatitis B or C).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-02; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Balo, Study Chair — DexCom, Inc.

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Clinical Research Centers during 12-Mar-2010 to 09-Apr-2010.
Pre-assignment Details: Prospective study- the investigator does not assign specific interventions to the subjects of the study in terms of their diabetes management.
Groups:
- Continuous Glucose Monitoring System: DexCom™ G4 Continuous Glucose Monitoring System : Continuous Glucose Monitoring System, that is a glucose monitoring device indicated for detecting trends and tracking patterns in persons with diabetes. The system is intended for single patient use and requires a prescription.
Period: Overall Study
Arm/Group | Continuous Glucose Monitoring System
Started | 60
Completed | 58
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- Continuous Glucose Monitoring System: The Dexcom G4 Continuous Glucose Monitoring System is a glucose monitoring device indicated for detecting trends and tracking patterns in persons with diabetes. The system is intended for single patient use and requires a prescription.
Arm/Group | Continuous Glucose Monitoring System
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 58
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 27
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: the Proportion of G4 CGM System in Agreement With the Reference Standard
Description: The proportion of G4 System values within (±) 20% of YSI reference value for glucose levels >80 mg/dL and (±) 20 mg/dL at YSI glucose levels <80 mg/dL. This is primarayly laboratory measurement outcome,and it is not measured by clinical outcome, for example, diagnosis, treatement and complication, and clinical effectiveness, etc.
Time Frame: Assessment done on either Day 1, 4 or 7 of the sensor wear period
Population: Randomly enrolled
Measure: Mean (95% Confidence Interval); unit: %20/20
Groups:
- CGM Device: DexCom™ G4 Continuous Glucose Monitoring System
Arm/Group | CGM Device
Number analyzed (Participants) | 60
%20/20 | 80 [78 to 82]

ADVERSE EVENTS:
Time Frame: 7 days
Groups:
- Real Time Continuous Glucose Monitoring System: continuous glucose monitoring system
  DexCom™ G4 Continuous Glucose Monitoring System: Continuous Glucose Monitoring System
Arm/Group | Real Time Continuous Glucose Monitoring System
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other